CLINICAL TRIAL: NCT02190760
Title: Comparison Between Perineural and Systemic Effect of Dexamethasone as an Adjuvant for Prolongation of the Interscalene Brachial Plexus Block.
Brief Title: Comparison Between Perineural and Systemic Effect of Dexamethasone for Interscalene Brachial Plexus Block.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HYMC-13.7.14
Record Dates: First submitted 2014-07-13; First posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Dexamethasone; Bupivacaine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group I (ISB-P) (Active Comparator): Interscalene block with perineural injection of dexamethasone 0.1 mg/kg
  Interventions: Drug: Dexamethasone; Drug: Bupivacaine
- Group II (ISB-S) (Active Comparator): Interscalene block with systemically injection of dexamethasone 0.1 mg/kg.
  Interventions: Drug: Dexamethasone; Drug: Bupivacaine
- Group III - ISB-C (Active Comparator): Interscalene block without adjuvant.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Dexamethasone
  Arms: Group I (ISB-P); Group II (ISB-S)
Drug: Bupivacaine

SUMMARY:
The addition of dexamethasone (DxaM) to local anesthetic may significantly prolong the duration of a block. The aim of this study is to determine whether this a systemic or local effect.

ELIGIBILITY:
Inclusion Criteria:

* Pre-surgical patients for arthroscopic or open shoulder surgery

Exclusion Criteria:

* Skin infection near block site
* Allergy to local anesthetics
* Peripheral neuropathy
* Proven opioid dependency
* Coagulopathy
* Dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy DxaM Perineural | One day
  Duration of motor and sensory block.

SECONDARY OUTCOMES:
Efficacy of Systemic DxaM | One day
  Duration of motor and sensory block

CONTACTS AND LOCATIONS:
Overall Officials: Anatoly Stav, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

REFERENCES:
- [Derived] Bei T, Liu J, Huang Q, Wu J, Zhao J. Perineural Versus Intravenous Dexamethasone for Brachial Plexus Block: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Pain Physician. 2021 Sep;24(6):E693-E707. PMID 34554686